CLINICAL TRIAL: NCT00334932
Title: Phase I/II Study of Liposomal Doxorubicin (Doxil®)/ Melphalan/Bortezomib (Velcade®) in Relapsed/Refractory Multiple Myeloma
Brief Title: Doxorubicin Hydrochloride Liposome, Melphalan, and Bortezomib in Treating Patients With Relapsed or Refractory Stage I, Stage II, or Stage III Multiple Myeloma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000471769; CPMC-AAAB6443
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2014-01-10 (Estimated); Status verified 2008-08

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bortezomib; Melphalan

INTERVENTIONS:
Drug: bortezomib
Drug: melphalan
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin hydrochloride liposome and melphalan, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving doxorubicin hydrochloride liposome and melphalan together with bortezomib may kill more cancer cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of doxorubicin hydrochloride liposome , melphalan, and bortezomib and to see how well they work in treating patients with relapsed or refractory stage I, stage II, or stage III multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and tolerability of doxorubicin HCl liposome, melphalan, and bortezomib in patients with relapsed or refractory stage I-III multiple myeloma.
* Determine the maximum tolerated dose (MTD) of this regimen in these patients.

Secondary

* Determine the overall response rate, including complete, near-complete, partial, and minimal response rate, in patients treated with this regimen.
* Determine the time to response, progression-free survival, and overall survival of patients treated with this regimen.
* Determine the toxic effects of this regimen at the MTD in these patients.

OUTLINE: This is a multicenter, phase I, dose-escalation study followed by a phase II study.

* Phase I: Patients receive doxorubicin HCl liposome IV over 30-60 minutes and melphalan IV over 30 minutes on day 1 and bortezomib IV on days 1, 4, 8, and 11. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of doxorubicin HCl liposome, melphalan, and bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 4 of 6 patients experience dose-limiting toxicity after 2 courses of therapy.

* Phase II: Patients receive doxorubicin HCl liposome, melphalan, and bortezomib at the MTD as in phase I.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: Approximately 32 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma

  * Stage I, II, or III disease according to Durie-Salmon staging criteria
* Progressive disease, defined as one of the following:

  * For secretory disease:

    * A 25% increase in serum M-protein or Bence Jones protein (an absolute increase of 0.5 g/dL serum M-protein or ≥ 200 mg/24 hours of urine light chain excretion)
  * For nonsecretory disease:

    * Bone marrow biopsy with > 25% increase in plasma cells or an absolute increase of ≥ 10% over prior known level
    * Development of new or worsening existing lytic bone lesions or soft tissue plasmacytomas
    * Hypercalcemia (i.e., calcium > 11.5 mg/dL)
    * Relapsed after complete response
* Must have received ≥ 2 of the following therapeutic regimens for multiple myeloma:

  * Nonmyeloablative transplantation

    * No significant graft-versus-host disease
    * At least 30 days since prior immunosuppressive therapy (concurrent prednisone allowed provided dose is ≤ 10 mg daily)
  * Mobilization with chemotherapy followed by either single or tandem autologous stem cell transplantation (considered 1 prior regimen)
  * Mobilization with chemotherapy followed by autologous and subsequent nonmyeloablative allogeneic stem cell transplantation (considered 1 prior regimen)
  * Any combination of drugs given concurrently (considered 1 prior regimen)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* Absolute neutrophil count > 1,000/mm^3 (no colony-stimulating factors)
* Platelet count > 50,000/mm^3 (no transfusion support)
* Bilirubin ≤ 2.0 mg/dL
* AST ≤ 4 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 4 weeks after completion of study treatment
* No history of allergic reaction to compounds containing boron or mannitol
* No active uncontrolled viral (including HIV), bacterial, or fungal infection
* No motor or sensory neuropathy ≥ grade 2
* No myocardial infarction within the past 6 months
* No New York Heart Association class III or IV heart failure
* No uncontrolled angina
* No severe uncontrolled arrhythmia
* No acute ischemia by EKG
* LVEF ≥ 35% by MUGA (MUGA required in patients whose lifetime cumulative doxorubicin hydrochloride dose > 400 mg/m^2)

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No grade III or IV toxicity due to previous antineoplastic therapy (except alopecia)
* At least 3 weeks since prior chemotherapy
* No prior doxorubicin HCl liposome, melphalan, and bortezomib as combination therapy (single or two-drug combinations of these are allowed)
* No concurrent corticosteroids (≤ 10 mg prednisone/day or equivalent allowed)
* No other concurrent chemotherapy
* No concurrent thalidomide
* No other concurrent investigational therapy
* No other concurrent antineoplastic treatment for multiple myeloma, including clarithromycin
* No concurrent radiation therapy
* No concurrent nonsteroidal anti-inflammatory agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2006-02; Primary Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients experiencing treatment-related ≥ grade 3 hematologic or nonhematologic toxicity or treatment-related death (phase I)

SECONDARY OUTCOMES:
Time to response (phase II)
Progression-free survival (phase II)
Overall survival (phase II)
Toxicities by NCI criteria (phase II)

CONTACTS AND LOCATIONS:
Overall Officials: Ajai Chari, MD, Principal Investigator — Herbert Irving Comprehensive Cancer Center
Locations (2):
- United States (2):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York

REFERENCES:
- [Result] Chari A, Kaplan L, Linker C, et al.: Phase I/II study of bortezomib in combination with liposomal doxorubicin and melphalan in relapsed or refractory multiple myeloma. [Abstract] Blood 106 (11): A-5182, 2005 .